CLINICAL TRIAL: NCT04298619
Title: Impact on Survival of Early Detection of Recurrence in the Follow Up of High Risk Hodgkin Lymphoma in First Complete Remission
Brief Title: Follow Up of High Risk Hodgkin Lymphoma in First Complete Remission
Acronym: HOLYFU
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Marco Picardi, Professor, Federico II University
Other Study IDs: HEM-FEDII-HL follow-up -001
Record Dates: First submitted 2020-03-03; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Hodgkin Lymphoma; High Risk; Relapse
MeSH Terms: conditions — Hodgkin Disease; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard cohort: Clinical-based surveillance after first complete remission in High risk Hodgkin Lymphoma patients:
  * symptom assessment
  * blood tests
  * physical examination
  Interventions: Diagnostic Test: Standard cohort: Clinical lab follow-up
- Imaging cohort: Clinical-based surveillance after first complete remission in High risk Hodgkin Lymphoma patients:
  * symptom assessment
  * blood tests
  * physical examination
  * Positron Emission Tomography (PET)/Computed Tomography (CT) or Chest X-Ray ultrasonography scan of superficial, mediastinal, abdominal and pelvic lymph nodes
  Interventions: Diagnostic Test: Standard cohort: Clinical lab follow-up; Diagnostic Test: Imaging cohort: integrated imaging follow-up

INTERVENTIONS:
Diagnostic Test: Standard cohort: Clinical lab follow-up
Diagnostic Test: Imaging cohort: integrated imaging follow-up
  Groups: Imaging cohort

SUMMARY:
Cohort study enrolled high-risk Hodgkin Lymphoma patients in first relapse after induction therapy followed after remission either with a systemic imaging-based surveillance (Imaging cohort) or with standard clinical-based surveillance (standard cohort).

ELIGIBILITY:
Inclusion Criteria:

* High risk Hodgkin Lymphoma
* achievement of complete response to first line therapy

Exclusion Criteria:

* comorbidities that could impair participation in follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Standard cohort: patients followed-up at the Santa Maria Loreto Mare Hospital Imaging cohort: patients followed-up at the University of Naples Federico II
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2001-06 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Event Free Survival (EFS) | Time period from the first relapse after induction therapy to the date of an event (refractoriness, relapse, or death) or the last follow-up visit after autologous stem cell transplantation (ASCT), up to 2 years
  Events:
  * refractoriness
  * relapse
  * death

SECONDARY OUTCOMES:
EFS for clinically silent relapses | Time period from the first relapse after induction therapy to the date of an event (refractoriness, relapse, or death) or the last follow-up visit after autologous stem cell transplantation (ASCT), up to 2 years
  Events:
  * refractoriness
  * relapse
  * death
Response rate | After salvage therapy and autologous stem cell transplantation (ASCT), up to 2 years
  Rate of response